CLINICAL TRIAL: NCT01709864
Title: A 12-week Multi-center, Randomized, Double-blind, Placebo Controlled Study to Assess the Efficacy and Safety of NVA237 in Stable COPD Patients
Brief Title: NVA237 Versus Placebo 12-week Efficacy Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNVA237A2317
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Anticholinergic; Antimuscarinic; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease; Chronic Obstructive Pulmonary Disease; COPD; LAMA; Lung Disease; Lung Diseases, Obstructive; Lung Function; Muscarinic receptor antagonist; Pulmonary Disease, Chronic Obstructive; Respiratory Tract Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Lung Diseases, Obstructive; Respiratory Tract Diseases | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVA237 (Experimental): NVA237 will be inhaled from a single-dose dry powder inhaler for a period of 12 weeks
  Interventions: Drug: NVA237
- Placebo (Placebo Comparator): Placebo will be inhaled from a single-dose dry powder inhaler for a period of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NVA237 — NVA237 (glycopyrronium bromide) as a powder for inhalation in single-dose capsules.
  Arms: NVA237
Drug: Placebo — Placebo powder for inhalation in single-dose capsules (matching those for NVA237).
  Arms: Placebo

SUMMARY:
The study serves to determine whether the treatment of patients with stable, symptomatic Chronic Obstructive Pulmonary Disease (COPD) with the investigational drug NVA237 is efficient and safe. The efficacy and safety of the drug will be tested against a placebo treatment.

The primary criterion to assess efficacy will be the difference between the serial lung function measurements of patients who have been treated for 12 weeks with NVA237 versus those that have received placebo treatment for 12 weeks. A serial lung function measurement (FEV1 testing) will be conducted and the "area under the curve" will be the measure for the ability to breathe.

ELIGIBILITY:
Inclusion criteria:

1. Patients with stable, symptomatic Chronic Obstructive Pulmonary Disease (COPD) with airflow obstruction of level 2 and 3 according to the current Global initiative for chronic Obstructive Lung Disease (GOLD) strategy (2011).
2. Patients with Forced Expiratory Volume in one second (FEV1) ≥ 30% and <80 % of the predicted normal, and FEV1/ Forced Vital Capacity (FVC) < 0.70 when measured 45 min after the inhalation of 84 µg ipratropium bromide.
3. Current or ex-smokers with at least 10 cigarette pack years smoking history.

Exclusion criteria:

1. Patients with a history of long QT syndrome, with a prolonged QTc measured during screening, or patients who have a clinically significant ECG abnormality at screening.
2. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
3. Pregnant or nursing (lactating) women. Women of childbearing potential unless using an effective method of contraception.
4. Patients who in the judgment of the investigator, would be at potential risk if enrolled into the study.
5. Patients who have a clinically significant concomitant disease at screening, including but not limited to clinically significant laboratory abnormalities, clinically significant renal, cardiovascular, neurological, endocrine, immunological, psychiatric, gastrointestinal, hepatic, or hematological abnormalities, or with uncontrolled diabetes, which could interfere with the assessment of the efficacy and safety of the study treatment.
6. Patients with a body mass index (BMI) of more than 40 kg/m2.
7. Patients contraindicated for treatment with, or having a history of reactions/ hypersensitivity to anticholinergic agents, long and short acting beta-2 agonists, or sympathomimetic amines.
8. Patients with any history of asthma, with onset of symptoms prior to age 40 years, or patients with a high blood eosinophil count during screening.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- United States (46):
  - Novartis Investigative Site, Homewood, Alabama
  - Novartis Investigative Site, Jasper, Alabama
  - Novartis Investigative Site, *See Various Dept.'s*, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Fountain Valley, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Brandon, Florida
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, DeFuniak Springs, Florida
  - Novartis Investigative Site, Edgewater, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Hialeah, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Pompano Beach, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, Summerfield, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Easley, South Carolina
  - Novartis Investigative Site, Gaffney, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Ninety Six, South Carolina
  - Novartis Investigative Site, Rock Hll, South Carolina
  - Novartis Investigative Site, Seneca, South Carolina
  - Novartis Investigative Site, Simpsonville, South Carolina
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Union, South Carolina
  - Novartis Investigative Site, Amarillo, Texas
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Beaumont, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Huntsville, Texas
  - Novartis Investigative Site, Waco, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NVA237 | Placebo
Started | 222 | 219
Full Analysis Set (FAS) | 222 (FAS included all randomized patients who received at least one dose of trial drug.) | 216 (FAS included all randomized patients who received at least one dose of trial drug.)
Per Protocol Set (PPS) | 204 (PPS included all patients in the FAS who did not have any major protocol deviations.) | 201 (PPS included all patients in the FAS who did not have any major protocol deviations.)
Completed | 215 | 208
Not Completed | 7 | 11
Not completed — Physician Decision | 0 | 1
Not completed — subject/guardian decision | 5 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — non-compliance with study treatment | 1 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVA237 | Placebo | Total
Number analyzed (Participants) | 222 | 219 | 441
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.36) | 62.1 (8.34) | 62.4 (8.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 87 | 185
  Male | 124 | 132 | 256

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Standardized Area Under the Curve (AUC) for Forced Expiratory Volume in One Second (FEV1) Post Dosing
Description: The standardized Area Under the Curve (AUC) for Forced Expiratory Volume in one second (FEV1) post dosing (FEV1 AUC) at week 12 of treatment. Serial lung function measurements are taken at various time points following dosing at week 12 to calculate the AUC.
Time Frame: 12 weeks
Population: The full analysis set (FAS): all randomized patients who received at least one dose of trial drug, patients were analyzed according to the treatment they were assigned to at randomization. analyzed participants had values at both baseline and the corresponding time frame, i.e. week 12
Measure: Least Squares Mean (Standard Error); unit: liters*hr
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 222 | 216
liters*hr | 0.125 (0.0162) | -0.014 (0.0165)

2. Secondary Outcome: Change From Baseline in Trough FEV1 and Pre-dose Trough FEV1 by Visit
Description: Trough Forced Expiratory Volume in one second (FEV1) is the mean of FEV1 at 23h 15min and 23h 45min after the morning dose of the previous day. Pre-dose trough FEV1 is the mean of FEV1 at -45min and -15min before morning dose
Time Frame: Day 2, 86 (trough) Day 15, 29, 57, 85 (pre-dose trough)
Population: The full analysis set (FAS): all randomized patients who received at least one dose of trial drug, patients were analyzed according to the treatment they were assigned to at randomization. However, for a given time frame, analyzed participants had values at both baseline and the corresponding time frame.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 222 | 216
liters
  Trough FEV1 Day 2 (n=218, n=214) | 0.141 (0.0124) | 0.025 (0.0122)
  Trough FEV1 Day 86 (n=218, n=214) | 0.123 (0.0171) | 0.007 (0.0173)
  Pre-dose Trough FEV1 Day 15 (n=217, n=208) | 0.112 (0.0135) | -0.002 (0.0135)
  Pre-dose Trough FEV1 Day 29 (n=217, n=208) | 0.0105 (0.0137) | -0.005 (0.0136)
  Pre-dose Trough FEV1 Day 57 (n=217, n=208) | 0.0106 (0.0156) | -0.006 (0.0157)
  Pre-dose Trough FEV1 Day 85 (n=217, n=208) | 0.090 (0.0155) | -0.029 (0.0157)

3. Secondary Outcome: Change From Baseline in FEV1 AUC (0-12H) at Day 1 and FEV1 AUC (0-4h), AUC (4-8h), AUC (8-12h) at Day 1 and Week 12 (Day 85)
Description: The standardized Area Under the Curve (AUC) for Forced Expiratory Volume in one second (FEV1) is assessed for different time spans within the overall serial measurement post dosing (FEV1 AUCs Time Spans), at day 1 and at week 12 of treatment. Serial lung function measurements are taken at various time points post dosing on day 1 and at week 12 to calculate the AUC for these different time spans.
Time Frame: Day 1 and Week 12 (Day 85)
Population: The full analysis set (FAS): all randomized patients who received at least one dose of trial drug, patients were analyzed according to the treatment they were assigned to at randomization. However, for a given time frame, analyzed participants had values at both baseline and the corresponding time frame, i.e. Day 1and Week 12
Measure: Least Squares Mean (Standard Error); unit: liters*hr
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 222 | 216
liters*hr
  FEV1, AUC 0-12h Day 1 (n=222, n=216) | 0.140 (0.0108) | -0.001 (0.0106)
  FEV1, AUC 0-4h Day 1 (n=222, n=216) | 0.174 (0.0103) | 0.021 (0.0101)
  FEV1, AUC 0-4h Day 85 (n=222, n=216) | 0.171 (0.0163) | 0.001 (0.0167)
  FEV1, AUC 4-8h Day 1 (n=222, n=215) | 0.138 (0.0123) | 0.001 (0.0121)
  FEV1, AUC 4-8h Day 85 (n=222, n=215) | 0.115 (0.0172) | -0.017 (0.0174)
  FEV1, AUC 8-12h Day 1 (n=222, n=215) | 0.102 (0.0122) | -0.037 (0.0120)
  FEV1, AUC 8-12h Day 85 (n=222, n=215) | 0.074 (0.0166) | -0.034 (0.0168)

4. Secondary Outcome: Change From Baseline in the Health Status Assessed by St. George's Respiratory Questionnaire
Description: The health status, as reported by the patients, is assessed using the St. George's Respiratory Questionnaire (SGRQ). The SGRQ is a 50 item scale assessing symptoms, patient activities and impact of the disease. Scores range from 0 to 100 units, with higher scores indicating more limitations. The assessment is based on total score as well as the percentage of patients with clinically significant improvement at week 12 versus day 1. A clinically meaningful improvement (MCID) in SGRQ is defined as a decrease of 4 or more units of the SGRQ scale in the total score, as compared to baseline (change from baseline).
Time Frame: Week 12
Population: The full analysis set (FAS): all randomized patients who received at least one dose of trial drug, patients were analyzed according to the treatment they were assigned to at randomization. However, for a given time frame, analyzed participants had values at both baseline and the corresponding time frame, i.e. Week 12
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 210 | 192
score | -4.4 (0.96) | -1.7 (0.96)

5. Secondary Outcome: Percentage of Participants With a Clinically Important Improvement of >=4units in the SGRQ Total Score at Week 12
Description: The health status, as reported by the patients, is assessed using the St. George's Respiratory Questionnaire (SGRQ). The assessment is based on total score as well as the percentage of patients with clinically significant improvement at week 12 versus day 1. A clinically significant improvement in SGRQ is defined as less than or equal to -4 change from baseline.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 210 | 192
percentage of participants | 49.0 | 40.6

6. Secondary Outcome: Breathlessness Assessed by Transition Dyspnea Index (TDI) Focal Score at Week 12
Description: Breathlessness at week 12 is measured using the Transition Dyspnea Index (TDI). On day 1, breathlessness is assessed by the Baseline Dyspnea Index (BDI). Patients are considered to have clinically significant improvement with the TDI score change versus BDI being equal to or greater than 1. TDI focal score is based on three domains: functional impairment, magnitude of task and magnitude of effort. Each domain is scored from -3 (major deterioration) to 3 (major improvement) to give an overall TDI focal score of -9 to 9. Higher numbers indicate a better score.
Time Frame: Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 200 | 188
scores on a scale | 1.46 (0.289) | 0.54 (0.286)

7. Secondary Outcome: Change From Baseline of Daily Symptom Scores
Description: Patients reported symptoms using an electronic diary.The diary has 9 symptom questions each am and each pm. Each question can be answered w/1 of 4 pre-defined answers, with a unit value of 0-3, 0 is least & 3 is most severe symptom.Symptom scores are calculated as the mean of combined daily symptom scores(combined from am & pm)for each patient over 12 weeks. The baseline is calculated from the run-in epoch prior to randomization.The change from baseline is in LS mean daily symptom scores over the 12 weeks. If the mean score over the 12 weeks is lower than the baseline, result is (-).A neg. result indicates an improvement in COPD symptom severity. Patients may have met the min. response requirements for the night scores(am questions),but not for the day scores(pm questions)or vice versa, the # of patients analyzed can vary between both day & night scores. Therefore, the # of patients analyzed for the combined daily symptom score can vary from the #s for individual day & night scores.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 211 | 204
Score | -1.39 (0.139) | -1.01 (0.135)

8. Secondary Outcome: Change From Baseline of Morning and Nighttime Symptom Scores at Week 12
Description: Patients reported symptoms using an electronic diary.The diary has 9 symptom questions each am & each pm.Each question can be answered w/1 of 4 pre-defined answers,with a unit value of 0-3, 0 is least & 3 is most severe symptom.Symptom scores are calculated as the mean of the symptom scores(either the score assessed in am for the previous 12 hrs-referred to as nighttime scores,or the score assessed in pm for the previous 12 hrs-referred to as the daytime symptom score) for each patient over 12 weeks.The baseline is calculated from the run-in epoch prior to randomization.The change from baseline is in LS mean daily symptom scores over the 12 weeks. If the mean score over the 12 weeks is lower than the baseline, result is (-).A neg. result indicates an improvement in COPD symptom severity. the # of patients analyzed can vary between both day & night scores. Therefore, the # of patients analyzed for the combined daily symptom score can vary from the #s for individual day & night scores.
Time Frame: 12 weeks
Population: Participants from the full analysis set (FAS), who had outcome measure data with applicable fixed effects/covariates according to the analysis model, were analyzed only and included all randomized patients who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 222 | 216
score
  Daytime total symptom score (n=208,202) | -1.14 (0.133) | -0.73 (0.130)
  nighttime total symptom score (n=207,202) | -1.22 (0.143) | -0.95 (0.139)

9. Secondary Outcome: Percentage of Nights With "no Nighttime Awakenings"
Description: Patients are reporting symptoms by using an electronic diary. A night with "no nighttime awakening" is defined from diary data as any night where the patient did not wake up due to symptoms. Percentage of no nighttime awakenings from Baseline up to 12 weeks.
Time Frame: from Baseline up to 12 weeks
Population: The full analysis set (FAS): all randomized patients who received at least one dose of trial drug. Following the intent-to -treat principle, patients were analyzed according to the treatment they were assigned to at randomization
Measure: Least Squares Mean (Standard Error); unit: percentage of nights
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 207 | 202
percentage of nights | 13.3 (2.00) | 11.3 (1.97)

10. Secondary Outcome: Percentage of Days With "no Daytime Symptoms"
Description: Patients are reporting symptoms by using an electronic diary. A day with "no daytime symptoms" is defined from diary data as any day where the patient has recorded in the evening no cough, no wheeze, no production of sputum, and no feeling of breathlessness (other than when running) during the past approximately 12 hours. The percentage of days is calculated by the number of days with no daytime symptoms/total number of days with evaluable data X 100.
Time Frame: from Baseline up to 12 weeks
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 208 | 202
percentage of days | 5.1 (1.65) | 2.5 (1.62)

11. Secondary Outcome: Percentage of "Days Able to Perform Usual Daily Activities"
Description: Patients are reporting symptoms by using an electronic diary. A "day able to perform usual daily activities" is defined from diary data as any day where the patient was not prevented from performing their usual daily activities due to respiratory symptoms.
Time Frame: from Baseline up to 12 weeks
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: pecentage of days
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 208 | 202
pecentage of days | 8.6 (2.20) | 1.8 (2.15)

12. Secondary Outcome: The Average Number of Puffs of Rescue Medication Per Day
Description: Patients report the number of puffs of rescue medication (salbutamol / albuterol) using an electronic diary. The use of rescue medication is analyzed as the mean daily number of puffs used per patient over the 12 weeks treatment period.
Time Frame: baseline and 12 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: number of puffs
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 211 | 204
number of puffs | -1.63 (0.180) | -0.86 (0.177)

13. Secondary Outcome: Percentage of Days Without Rescue Medication Use
Description: Patients report the number of puffs of rescue medication (salbutamol / albuterol) using an electronic diary. The use of rescue medication is analyzed as the percentage of days without usage of rescue medication over the 12 weeks treatment period. The baseline is calculated from the run-in epoch prior to randomization.
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 209 | 202
percentage of days | 16.6 (2.37) | 10.5 (2.31)

14. Secondary Outcome: Change From Baseline of Forced Vital Capacity (FVC) at All Individual Timepoints at Day 1 and at Week 12 (Day 85)
Description: The Forced Vital Capacity (FVC) assessments for all individual time points of the serial measurements on day 1 and at week 12 are analyzed.
Time Frame: Baseline, Day 1 and Week 12 (Day 85)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 222 | 216
liters
  DAY 1/ 5 min (n=221, 214) | 0.175 (0.0152) | 0.037 (0.0152)
  DAY 1/ 15 min (n=222, 216) | 0.265 (0.0181) | 0.044 (0.0180)
  DAY 1/ 1h (n=222, 216) | 0.318 (0.0207) | 0.032 (0.0205)
  DAY 1/ 2h (n=221, 216) | 0.351 (0.0216) | 0.071 (0.0213)
  DAY 1/ 4h (n=220, 213) | 0.290 (0.0235) | 0.067 (0.0231)
  DAY 1/ 6h (n=221, 214) | 0.252 (0.0235) | 0.022 (0.0234)
  DAY 1/ 8h (n=220, 214) | 0.192 (0.0221) | -0.009 (0.0220)
  DAY 1/ 11h 55min (n=216, 207) | 0.152 (0.0234) | -0.030 (0.0235)
  DAY 85/ -45 min (n=217, 208) | 0.162 (0.0289) | -0.043 (0.0296)
  DAY 85/ -15 min (n=216, 208) | 0.156 (0.0283) | -0.017 (0.0287)
  DAY 85/ 5 min (n=221, 214) | 0.184 (0.0282) | -0.007 (0.0287)
  DAY 85/ 15 min (n=222, 216) | 0.263 (0.0288) | -0.003 (0.0294)
  DAY 85/ 1h (n=222, 216) | 0.258 (0.0297) | 0.004 (0.0302)
  DAY 85/ 2h (n=221, 216) | 0.277 (0.0299) | 0.033 (0.0307)
  DAY 85/ 4h (n=220, 213) | 0.215 (0.0317) | 0.076 (0.0321)
  DAY 85/ 6h (n=221, 214) | 0.199 (0.0304) | -0.015 (0.0305)
  DAY 85/ 8h (n=220, 214) | 0.128 (0.0303) | -0.023 (0.0305)
  DAY 85/ 11h 55min (n=216, 207) | 0.110 (0.0286) | -0.006 (0.0288)

15. Secondary Outcome: Change From Baseline of Forced Expiratory Volume in One Second (FEV1) at All Individual Timepoints at Day 1 and at Week 12 (Day 85)
Description: The Forced Expiratory Volume in one second (FEV1) assessments for all individual time points of the serial measurements on day 1 and at week 12 are analyzed.
Time Frame: Baseline, Day 1 and Week 12 (Day 85)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 222 | 216
liters
  DAY 1/ 5 min (n=221, 214) | 0.074 (0.0075) | 0.015 (0.0074)
  DAY 1/ 15 min (n=222, 216) | 0.129 (0.0085) | 0.015 (0.0084)
  DAY 1/ 1h (n=222, 216) | 0.176 (0.0108) | 0.008 (0.0106)
  DAY 1/ 2h (n=221, 216) | 0.198 (0.0120) | 0.031 (0.0118)
  DAY 1/ 4h (n=220, 213) | 0.168 (0.0132) | 0.028 (0.0129)
  DAY 1/ 6h (n=221, 214) | 0.132 (0.0135) | 0.000 (0.0134)
  DAY 1/ 8h (n=220, 214) | 0.113 (0.0129) | -0.022 (0.0128)
  DAY 1/ 11h 55min (n=216, 207) | 0.083 (0.0131) | -0.046 (0.0131)
  DAY 85/ -45 min (n=217, 208) | 0.092 (0.0154) | -0.040 (0.0158)
  DAY 85/ -15 min (n=216, 208) | 0.090 (0.0160) | -0.022 (0.0162)
  DAY 85/ 5 min (n=221, 214) | 0.118 (0.0161) | -0.018 (0.0163)
  DAY 85/ 15 min (n=222, 216) | 0.171 (0.0164) | -0.016 (0.0168)
  DAY 85/ 1h (n=222, 216) | 0.178 (0.0166) | -0.014 (0.0169)
  DAY 85/ 2h (n=221, 216) | 0.186 (0.0178) | 0.006 (0.0183)
  DAY 85/ 4h (n=220, 213) | 0.147 (0.0180) | 0.014 (0.0182)
  DAY 85/ 6h (n=221, 214) | 0.120 (0.0183) | -0.026 (0.0183)
  DAY 85/ 8h (n=220, 214) | 0.080 (0.0180) | -0.036 (0.0181)
  DAY 85/ 11h 55min (n=216, 207) | 0.072 (0.0165) | -0.043 (0.0165)

ADVERSE EVENTS:
Arm/Group | NVA237 | Placebo
Serious Adverse Events (participants affected / at risk) | 11/222 | 12/216
Other Adverse Events (participants affected / at risk) | 72/222 | 66/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=222) | Placebo (N=216)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 2
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 1
WOUND INFECTION (Infections and infestations) | 0 | 1
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 1 | 0
HEAT STROKE (Injury, poisoning and procedural complications) | 1 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
VOLUME BLOOD DECREASED (Investigations) | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 0.9% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=222) | Placebo (N=216)
VERTIGO (Ear and labyrinth disorders) | 3 | 0
VISION BLURRED (Eye disorders) | 2 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 3
DIARRHOEA (Gastrointestinal disorders) | 2 | 2
DRY MOUTH (Gastrointestinal disorders) | 1 | 2
NAUSEA (Gastrointestinal disorders) | 1 | 2
FATIGUE (General disorders) | 0 | 2
OEDEMA PERIPHERAL (General disorders) | 2 | 2
BRONCHITIS (Infections and infestations) | 3 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 2
INFLUENZA (Infections and infestations) | 2 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 0
NASOPHARYNGITIS (Infections and infestations) | 3 | 7
ORAL CANDIDIASIS (Infections and infestations) | 2 | 1
PNEUMONIA (Infections and infestations) | 3 | 0
SINUSITIS (Infections and infestations) | 3 | 2
TOOTH ABSCESS (Infections and infestations) | 0 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 | 6
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 2 | 4
URINARY TRACT INFECTION (Infections and infestations) | 3 | 3
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 3
EXCORIATION (Injury, poisoning and procedural complications) | 2 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 0
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1
DIZZINESS (Nervous system disorders) | 0 | 2
HEADACHE (Nervous system disorders) | 8 | 6
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 2
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 22 | 26
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 | 4
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 4
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2
HYPERTENSION (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.